CLINICAL TRIAL: NCT05189873
Title: Comparison of the Pregnancy Outcomes in Patients With the Polycystic Ovarian Syndrome in Two Endometrial Preparation Method GnRH Agonist Plus Hormone Replacement Therapy Versus Hormone Replacement Therapy in Frozen Embryo Transfer Cycle
Brief Title: GnRH Agonist Plus Hormone Replacement Therapy vs Hormone Replacement Therapy on IVF Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-3-101-51284
Record Dates: First submitted 2021-12-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Polycystic Ovary Syndrome; Infertility, Female
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization list will be prepared by a statistician using the block randomization method (using the site:www.sealedenvelope.com). Treatments are placed in sealed envelopes and will be kept by the out-of-study nurse. After identification of the eligibility of the patient, the procedure is explained to her and informed consent is obtained. Then the treatment is performed based on the kind of treatment in the envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRT (Experimental): HRT protocol : estradiol and progesterone
  Interventions: Drug: HRT
- Long GnRH agonist + HRT (Experimental): Long GnRH agonist + HRT protocol: Superfect and estradiol and progesterone
  Interventions: Drug: Long GnRH agonist + HRT

INTERVENTIONS:
Drug: Long GnRH agonist + HRT — Intervention group:(Long GnRH agonist + HRT) From day 18-21 of the previous cycle, 0.5 cc of Superfect is injected daily and vaginal ultrasound is performed 10-14 days later If the endometrial thickness is less than 5 mm and there are no ovarian cysts, estradiol is started like HRT treatment and the agonist dose of GnRH starts with estradiol. It is halved (0.25 cc superfect) and superfect is prescribed until progesterone is started. At the time of progesterone administration, the administration of superfect is discontinued. Injections of estradiol and progesterone is the same as for the HRT group
  Arms: Long GnRH agonist + HRT
Drug: HRT — In the HRT group, from the second day of the cycle, the participant receives 2 mg of estradiol daily and this drug is increased to 6 mg per day in three days.Ten days later, they undergo vaginal ultrasound to check the thickness of the endometrium. If the thickness of the endometrium is greater than 8 mm, inject able progesterone is prescribed and the patient is a candidate for FET transfer. If the thickness is less than 7 mm, it is necessary to increase the dose of estradiol and continue treatment with it. The patient undergoes vaginal ultrasound every three days and if the desired thickness does not reach 21 days after the start of the cycle, the cycle is canceled
  Arms: HRT

SUMMARY:
The study is conducted at Arash Women's Hospital on all women undergoing the frozen embryo transfer cycle. Patients who signed informed consent will be randomly divided into two groups. The first group will receive GnRH agonist plus hormone replacement therapy for endometrial preparation. Group 2 will receive hormone replacement therapy. The random allocation and final outcome of the study will be assessed by a person who is unaware of the study process. Also, the statistician will be unaware of the study process

ELIGIBILITY:
Inclusion Criteria:

The first or second cycle of embryo transfer Normal uterine cavity PCO diagnosis based on Rotterdam criteria and correction (2018) Age 20 to 40 years

Exclusion Criteria:

Infertility with severe male factor endometriosis immunological disease FSH higher than 10 BMI greater than or equal to 30 Endometrial thickness on the day of transfer is less than 7 mm History of recurrent miscarriage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | On the day of transfer
  Endometrial thickness on the day of transfer will be measured by transvaginal ultrasound
Chemical pregnancy | 14 days after transfer
  A positive beta hCG levels
Clinical pregnancy | 12 weeks of pregnancy
  The gestational sac will be observed by Ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Moini, professor, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Arash women's hospital,Tehran university of medical sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make this available